CLINICAL TRIAL: NCT06851416
Title: Cross-Cultural Adaptation and Psychometric Evaluation of the Critical Care Pressure Ulcer Assessment Tool Made Easy (CALCULATE) in a Critical Care Unit in Turkey
Brief Title: Cross-Cultural Adaptation on CALCULATE in a Critical Care Unit
Acronym: CALCULATE
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cansu POLAT DÜNYA, Asisst Prof, Istanbul University
Other Study IDs: 28.08.2024 /2024-353
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pressure Injury; Critical Care
Keywords: pressure injury; critical care; validity; reliability
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patient: Patients who are 18 years or older, without a pressure injury at the time of ICU admission, expected to stay in the ICU for at least 72 hours, and who consent to participate in the study (or whose family members consent) included in the study. Patients or their family members who did not consent to participate, as well as patients who transferred to another hospital during their ICU stay, excluded from the study.

SUMMARY:
Pressure injuries are localized lesions that occur in the skin and/or underlying tissues due to pressure, or pressure in combination with shear. PIs arise as a consequence of prolonged immobility during hospitalization, leading to increased morbidity, mortality, prolonged hospital stays which may result in higher healthcare costs. Critically ill patients are vulnerable cohort of patients at a higher risk of developing PIs compared to the general population due to factors such as immobility, severity of illness, hemodynamic instability, ventilation, use of vasopressors, and the application of medical devices.

DETAILED DESCRIPTION:
Despite the potential for preventing pressure injury through evidence-based, multidisciplinary approaches, critically ill patients still develop pressure injury at approximately four times the rate of other patients.While there are over forty pressure injuries risk assessment tools available, none are considered the 'gold standard,' and their assessments are based on subjective data, which may not yield valid and reliable results in clinical practice. In a study identified sixteen scales used to assess pressure injury in intensive care, with the Cubbin and Jackson Index, Braden, and Waterlow being the most common. Although the Braden scale was most frequently used, it was not considered the best tool for intensive care unit patients. In a recent review, the Critical Care Pressure Ulcer Assessment Tool made Easy was noted to outperform others in detecting pressure injuries, with the Braden and Critical Care Pressure Ulcer Assessment Tool made Easy scores showing superior performance, and Braden demonstrating the best results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older
* without a pressure injury at the time of ICU admission
* expected to stay in the ICU for at least 72 hours
* who consent to participate in the study (or whose family members consent) included in the study.

Exclusion Criteria:

* Patients or their family members who did not consent to participate,
* Patients who transferred to another hospital during their ICU stay, excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patient
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
CALCULATE Pressure Ulcer Risk Assessment Scale in Intensive Care | 3 days
  The CALCULATE was developed by Richardson and Straughan (2015) to evaluate the risk of pressure ulcer development in intensive care patients. The scale was later revised and published in its final form by Richardson and Straughan (2015), consisting of eight items. These items assess eight pressure ulcer risk factors: mechanical ventilation, impaired circulation, dialysis, prolonged surgery/cardiac arrest (surgery duration> 4 hours in the last 24 hours or cardiac arrest during this hospital stay), fecal incontinence (diarrhea type 5, 6, or 7), low protein (albumin <35 g/L and/or malnutrition), immobility, and instability to the extent that the patient cannot turn. Each risk factor is assigned one point, with the total score ranging from 0 to 8. Based on the scoring, patients with four or more risk factors are classified as "very high risk," while those with three or fewer risk factors are classified as "high risk."

SECONDARY OUTCOMES:
Braden Pressure Ulcer Risk Assessment Scale | 3 days
  The Braden Pressure Ulcer Risk Assessment Scale, developed by Braden and Bergstrom (1987), was adapted into Turkish by Karadag and Avşar (2013). The scale consists of six subscales: sensory perception, moisture, activity, mobility, nutrition, and friction and shear. The subscales of sensory perception, moisture, activity, mobility, and nutrition are scored between 1 and 4, while the friction and shear subscale is scored between 1 and 3. The total score on the scale ranges from a minimum of 6 to a maximum of 23. Lower scores indicate a higher risk of developing a pressure ulcer . A total score of 15-16 indicates a low risk, 13-14 indicates a moderate risk, and 12 or below indicates a high risk. For patients aged 75 and older, a score of 15-18 is considered low risk
Biochemical Markers | 1 day
  Based on the literature (Hatanaka et al., 2008; Wang et al., 2022), albumin, hemoglobin, and CRP levels monitored daily throughout the patient's stay in the intensive care unit. In the intensive care unit where the study conducted, these biochemical markers are routinely measured daily for all ICU patients

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Özen, Assoc. Prof, RN, PhD, Principal Investigator — Istanbul University, Istanbul, Turkey; Fatma Nur Ceylan, MScN, Study Chair — Isparta City Hospital, Isparta, Turkey; Aysegül Ünlü, Study Chair — Isparta City Hospital, Isparta, Turkey; Natalie McEvoy, RN, PhD, Study Chair — Royal College of Surgeons, Ireland
Locations (1):
- Istanbul University, Fatih, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Theeranut A, Ninbanphot S, Limpawattana P. Comparison of four pressure ulcer risk assessment tools in critically ill patients. Nurs Crit Care. 2021 Jan;26(1):48-54. doi: 10.1111/nicc.12511. Epub 2020 May 5. PMID 32368844
- [Result] Richardson A, Straughan C. Part 2: pressure ulcer assessment: implementation and revision of CALCULATE. Nurs Crit Care. 2015 Nov;20(6):315-21. doi: 10.1111/nicc.12172. Epub 2015 Mar 19. PMID 25787803